CLINICAL TRIAL: NCT06561802
Title: Evaluation Of Gingival Crevicular Fluid And Salivary Ferritin, Alkaline Phosphatase And Matrix Metalloproteinase-8 Levels Of Individuals With Different Periodontal Diseases
Brief Title: Evaluation of GCF And Salivary Ferritin, ALP And MMP-8 Levels of Individuals With Different Periodontal Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Erim Bozkurt, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-TDR-SABE-0009
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periodontally healthy (Experimental): Full-mouth clinical periodontal measurements recorded and GCF and saliva obtained.
  Interventions: Diagnostic Test: GCF and saliva obtaining
- gingivitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF and saliva obtained.
  Interventions: Diagnostic Test: GCF and saliva obtaining
- periodontitis (Experimental): Full-mouth clinical periodontal measurements recorded and GCF and saliva obtained.
  Interventions: Diagnostic Test: GCF and saliva obtaining

INTERVENTIONS:
Diagnostic Test: GCF and saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Also, 4 samples of gingival crevicular fluid, 1 from each quadrant of the patient's jaw, were collected by means of paper strips and put into propylene tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
The aim of this clinical study was to determine the levels of ferritin, alkaline phosphatase and matrix metalloproteinase-8 in the gingival crevicular fluid (GCF) and saliva samples were collected from 60 systemically healthy, non-smoker periodontitis (P group, n = 20), gingivitis (G group, n = 20) and periodontally healthy individuals (S group, n = 20) and all clinical parameters were recorded for all groups at baseline. GCF and serum samplings and clinical records were also repeated at 1st and 3rd months visitsfor only P group. Ferritin, MMP8, and ALP levels in samples were determined by enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* At least twenty permanent teeth in the mouth
* Non-smoker
* No medication for continuous use
* Those who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months.
* Not in pregnancy or lactation period.
* For the periodontitis group that has not received periodontal treatment in the last 6 months

  * For the periodontitis group; According to the evaluation made in 6 regions of each tooth, individuals with 30% or more bleeding on probing area, at least 2 teeth not adjacent to each quarter jaw with a depth of 5 mm or more and 4 mm or more attachment loss, coronal 1/3 and more on radiography (horizontal and / or vertical) bone loss
  * For the gingivitis group; According to the evaluation made in 6 regions of each tooth, individuals with 10% or more bleeding on probing area, having a probing depth of less than 4mm and no attachment loss
  * For healthy group; According to the evaluation made in 6 regions of each tooth,individuals with less than 10% bleeding on probing area, having a probing depth less than 4mm and no loss of attachment were included in the study.

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months
* Smokers are not included in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The total amount of Ferritin in GCF and saliva | 24 hours after taking the clinical measurements at the first visit
The total amount of ALP in GCF and saliva | 24 hours after taking the clinical measurements at the first visit

SECONDARY OUTCOMES:
The total amount of MMP-8 in GCF and saliva | 24 hours after taking the clinical measurements at the first visit

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF